CLINICAL TRIAL: NCT04647539
Title: Emerging Invasive Fungal Infections in Critically Ill Patients: Epidemiological Trends, Clinical Features and Outcomes
Brief Title: Emerging Invasive Fungal Infections in Critically Ill Patients
Acronym: EIFI
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0626
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Fungal Infection; ICU Acquired Weakness
Keywords: Emergind invasive fungal infection; mucormycosis; ICU
MeSH Terms: conditions — Mycoses; Mucormycosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — NC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: Beside Candida and Aspergillus, emerging invasive fungal infections (EIFIs) are increasing in intensive care setting and are associated with high morbidity and mortality. However, data are scarce, particularly in ICU settings and for EIFIs other than mucormycosis.

Objectives: to describe epidemiological trends and clinical features of EIFIs in intensive care units (ICU) and to assess their outcome.

Methods: All records of adult patients diagnosed with an EIFI in a medical ICU between 2006 and 2019 were analyzed retrospectively. In-ICU mortality was assessed, then factors associated with mortality were identified. Survival at day-90 was calculated by the Kaplan-Meier method.

ELIGIBILITY:
Inclusion criteria:

- Adults (≥ 18 years old) with at least 1 positive culture for molds other than candida and aspergillosis

Exclusion criteria:

- Age < 18, pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients majeurs hospitalisés en reanimation et présentant une infection fongique invasive autre qu'une candidose ou une aspergilloses
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
mortality | at ICU admission
  mortality

SECONDARY OUTCOMES:
Mucormycosis | at ICU admission
  Mucormycosis

CONTACTS AND LOCATIONS:
Overall Officials: Romaric Larcher, MD, PharmD, MSc, Principal Investigator — UH Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC